CLINICAL TRIAL: NCT02299232
Title: Comparison of Two Different Intranasal Doses of Dexmedetomidine in Children for Magnetic Resonance Imaging (MRI) Sedation
Brief Title: Dexmedetomidine in Children for Magnetic Resonance Imaging (MRI) Sedation
Acronym: DEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Canan Tulay ISIL, M.D., Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 295/25.02.2014
Record Dates: First submitted 2014-11-05; First posted 2014-11-24 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Anesthesia
Keywords: dexmedetomidine; sedation; MRI
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine 3mcg/kg (Active Comparator): dexmedetomidine 3 mcg/kg intranasal 50 minutes before MRI
  Interventions: Drug: Dexmedetomidine
- dexmedetomidine 4mcg/kg (Active Comparator): dexmedetomidine 4 mcg/kg intranasal 50 minutes before MRI
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Drug: dexmedetomidine 100 mcg/mL was applied in 3 mcg/kg and 4 mcg/kg doses in 1 mL preperates, 0.5 mL for each nostril
  Other Names: precedex

SUMMARY:
Sixty patients aged between 1-10 years, American Society of Anesthesia (ASA) physical status I-II scheduled for MRI were allocated in this randomized double-blinded study. Group 1 received 3 mcg/kg, Group 2 received 4 mcg/kg intranasal dexmedetomidine before imaging. From the beginning on every 10 minutes heart rate (HR), saturation (SpO2) and Ramsey Sedation Score (RSS) were recorded. Induction time was time interval to receive RSS 5. MRI began and separation-score was noted. If intranasal sedation failed, an intravenous canula was placed and propofol was applied. Imaging quality was evaluated. Recovery time was time interval to receive Aldrete-score 9. Parents' satisfaction was questioned before patient was discharged.

DETAILED DESCRIPTION:
OBJECTIVES OF STUDY Anesthetic agents used for MRI in paediatrics should have few adverse effects, allow fast induction and recovery. The administration route is also important and should be minimally invasive. In this study the investigators aimed to compare two different doses of intranasal dexmedetomidine applied to children for MRI sedation.

MATERIALS AND METHODS Sixty patients aged between 1-10 years, ASA I-II scheduled for MRI were allocated in this randomized double-blinded study. Group 1 received 3 mcg/kg, Group 2 received 4 mcg/kg intranasal dexmedetomidine before imaging. From the beginning on every 10 minutes HR, SpO2 and RSS were recorded. Induction time was time interval to receive RSS 5. MRI began and separation-score was noted. If intranasal sedation failed, an intravenous canula was placed and propofol was applied. Imaging quality was evaluated. Recovery time was time interval to receive Aldrete-score 9. Parents' satisfaction was questioned before patient was discharged.

ELIGIBILITY:
Inclusion Criteria:

* MRI
* ASA I-II

Exclusion Criteria:

* hepatic and renal failure
* difficult airway
* nasal deformity
* anaphylaxis to dexmedetomidine
* neurologic disease
* metabolic disorders
* electrolyte imbalance
* dehydration
* malnutrition

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Ramsey Sedation Score | every 10 minutes for a two hours period
  a score to determine sedation deepness

CONTACTS AND LOCATIONS:
Overall Officials: Hacer Sebnem Turk, MD, Principal Investigator — Sisli Hamidiye Etfal Training and Research Hospital

REFERENCES:
- [Background] Ambi US, Joshi C, Ganeshnavar A, Adarsh E. Intranasal dexmedetomidine for paediatric sedation for diagnostic magnetic resonance imaging studies. Indian J Anaesth. 2012 Nov;56(6):587-8. doi: 10.4103/0019-5049.104588. No abstract available. PMID 23325950
- [Background] Gyanesh P, Haldar R, Srivastava D, Agrawal PM, Tiwari AK, Singh PK. Comparison between intranasal dexmedetomidine and intranasal ketamine as premedication for procedural sedation in children undergoing MRI: a double-blind, randomized, placebo-controlled trial. J Anesth. 2014 Feb;28(1):12-8. doi: 10.1007/s00540-013-1657-x. Epub 2013 Jun 26. PMID 23800984
- [Derived] Tug A, Hanci A, Turk HS, Aybey F, Isil CT, Sayin P, Oba S. Comparison of Two Different Intranasal Doses of Dexmedetomidine in Children for Magnetic Resonance Imaging Sedation. Paediatr Drugs. 2015 Dec;17(6):479-85. doi: 10.1007/s40272-015-0145-1. PMID 26323489